CLINICAL TRIAL: NCT04817098
Title: Journey of Life Psychosocial Support for Conflict-Affected Populations in Uganda
Brief Title: Journey of Life Psychosocial Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: TPO Uganda (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 202101122
Record Dates: First submitted 2021-02-12; First posted 2021-03-25 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Psychological; Child Development; Social Values
Keywords: Refugee; Community development

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Journey of Life Intervention Group (Experimental): Community members (caregivers, teachers, and community leaders) will participate in group workshops for a period of 6 weeks.
  Interventions: Behavioral: Journey of Life
- Waitlist Control Group (Other): The waitlist control group will not receive the intervention during the first 6 months of implementation in order to assess the effects of the intervention compared to the control group. However, following intervention completion in the experimental group, the control group will receive 6 months of the intervention.
  Interventions: Behavioral: Journey of Life

INTERVENTIONS:
Behavioral: Journey of Life — The concept underlying the JoL intervention is that caregivers and community members can support each other and their children through reflection, dialogue, and action. JoL addresses children's and adolescents' ecologies by working with caregivers, educators, and community members to understand the importance of their support in protecting children.

SUMMARY:
The proposed study evaluates the impact and implementation of the Journey of Life intervention among crisis-affected caregivers living in Western Uganda. In this quasi experimental waitlist control design, participants will be assigned to treatment or waitlist control group based on their geographic location. The intervention will be delivered in X sessions weekly. Assessments will be conducted at baseline and following the intervention period. Assessments will include mental health, functioning, social support, child protection behaviors, parenting attitudes, and experiences of intimate partner violence. The study also aims to examine implementation of the Journey of Life intervention through qualitative assessments of feasibility, acceptability, adaptation, reach, and adoption.

DETAILED DESCRIPTION:
Aligned with the USAID HEARD (Health Evaluation and Applied Research Development) purpose to leverage global partnerships to generate, synthesize, and use evidence to improve program implementation in low and middle-income countries, the proposed study will examine the impact and implementation of the Journey of Life (JoL) intervention in a humanitarian setting. The JoL intervention aims to provide psychosocial support to adults and galvanize caregivers to develop action plans for child protection in their communities. The proposed research will involve an analysis of effect sizes for mental health, functioning, social support, child protection behaviors, parenting attitudes and behaviors, and experiences of intimate partner violence. The research also aims to interrogate implementation strategies that are useful within humanitarian contexts through qualitative key informant interviews and focus group discussions. Assessments include baseline and follow up data collection to measure effect sizes and assess implementation strategy components. The study aims are to: (1) assess the impact of JoL on child protection indicators, (2) examine the effects of JoL on behavioral health functioning (i.e. mental health, social support, and functioning)

ELIGIBILITY:
Inclusion Criteria:

* Refugee living in Kiryandongo settlement
* Over the age of 18
* Caregiver for a child under age 18

Exclusion Criteria:

* Anyone aged 17 and under, unless written consent from the caregiver and assent from the participant is provided
* Anyone unable to provide consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Mental health | 6 months
  Changes in mental health symptoms according to the Kessler-6 from baseline to follow up assessments. The structure of the survey asks participants how frequently they have experienced certain symptoms in the past thirty days and presents a consistent scale of responses ranging from "1 - All of the time" to "5 - None of the time"

SECONDARY OUTCOMES:
Functioning | 6 months
  Changes in functioning according to the World Health Organization Disability Assessment Schedule (WHODAS) from baseline to follow up. The WHODAS uses a 12-item scale with a range of scores from 12 to 60, where higher scores indicate higher disability or loss of function.
Social support | 6 months
  Changes in social supports according to the Medical Outcomes Study Social Supports 8-item survey from baseline to follow up. The survey is scored using an average of scores for each item and transferring them to a 0-100 score where a higher score for an individual indicates more support.
Child protection attitudes | 6 months
  Changes in the adoption of positive child protective behaviors from baseline to follow-up assessments according to the adapted Child Protection Index (CPI). The CPI is a 12-item instrument that assesses attitudes towards child protection with a scoring range of 0-12 wherein a higher number indicates more permissible attitudes towards beating children.
Parenting behaviors | 6 months
  Changes in the adoption of positive parenting behaviors from baseline to follow-up assessments according to the Parenting Acceptance and Rejection Questionnaire (PARQ). This 12-item subscale has a scoring range of 0-48 wherein higher scores indicate more acceptance of children.

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - TPO Uganda, Bweyale
  - TPO Uganda, Kiryandongo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen F, Hermosilla S, Knox J, Agaba GS, Obalim G, Kajungu R, Mangen PO, Stark L. Protocol for a caregiver psychosocial support intervention for populations affected by displacement in Uganda. BMC Public Health. 2021 May 17;21(1):932. doi: 10.1186/s12889-021-10921-7. PMID 34001055